CLINICAL TRIAL: NCT00430482
Title: Stress, Distress Intolerance, and Drug Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Michael Otto, Ph.D., Boston University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01DA017904 (NIH); R01DA017904 (NIH)
Record Dates: First submitted 2007-01-31; First posted 2007-02-02 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Substance Dependence
Keywords: Substance Dependence; Cognitive-Behavior Therapy; Opiate Dependence; Treatment Moderators
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Cognitive Behavioral Therapy
  Interventions: Behavioral: Cognitive Behavioral Therapy
- 2 (Active Comparator): Individual Counseling
  Interventions: Behavioral: Individual Counseling

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — 12 weekly sessions and 3 booster sessions of cognitive behavioral therapy
  Other Names: CBT
  Arms: 1
Behavioral: Individual Counseling — 12 weekly sessions and 3 booster sessions of individual counseling
  Other Names: ICT
  Arms: 2

SUMMARY:
This study is designed to evaluate the relative efficacy of a novel treatment (CBT-IC) versus a standard individual drug-counseling treatment. The novel treatment emphasizes exposure to emotional cues for drug use as part of a comprehensive, yet brief, treatment strategy. These treatments are delivered to opiate-dependent, often poly-substance dependent, individuals in a comprehensive methadone maintenance program who have failed to respond adequately to current treatments.

DETAILED DESCRIPTION:
This study study is designed to test further the efficacy of Cognitive-Behavior Therapy for Interoceptive Cues (CBT-IC - a treatment with a central focus on enhancing a patient's tolerance to the myriad forms of distress-sadness, boredom, anxiety, withdrawal sensations, etc.-that are linked to the stressful lives of drug-dependent individuals, and breaking the link between these emotional cues and drug-related attempts to avoid emotional distress) for intervening with chronically-stressed and treatment-resistant opiate-dependent outpatients. Features of this study of particular relevance to to RFA DA-04-001 include: (1) a focus on opiate-dependent patients undergoing chronic stress; (2) a model for the way in which chronic stress translates into chronic drug use; (2) a focus on the way in which stress-related symptoms serve as trigger for drug use; (3) a focus on both mediators and moderators of treatment that will inform treatment-matching efforts, including a focus on gender differences and emotional avoidance/distress intolerance; and (4) the examination of treatment outcome in a Stage II treatment trial.

ELIGIBILITY:
Inclusion Criteria:

* The primary selection criteria include women and men between the ages of 18 and 65 who:

  1. Meet DSM-IV criteria for opiate dependence,
  2. Maintain a stable dose of methadone for two weeks prior to recruitment and,
  3. a) fail to achieve "take-home" status for methadone dosing during at least the first four months of methadone treatment, b) test positive on at least two toxicology screens for illicit drugs during the month prior to recruitment c) have never achieved two consecutive toxicology screens free of illicit substances since entering the current treatment episode.
  4. Meet study criteria for chronic stress

     1. unemployment criteria, and
     2. affective disorder criteria.

Exclusion Criteria:

* (1) Patients with significantly unstable or uncontrolled medical illness which may interfere with participation in treatment (e.g., patients likely to require hospitalization during the study period).

  (2) Patients with a psychotic or organic mental disorder according to DSM-IV criteria.

  (3) Patients receiving medication affecting methadone metabolism (e.g. rifampin).

  (4) Patients with uncontrolled bipolar disorder as evidenced by meeting current criteria for mania or hypomania or meeting criteria for rapid cycling in the last year (as indicated by structured questioning of all patients meeting criteria for bipolar disorder).

  (5) Patients unable to complete the informed consent or unable to understand study procedures in the informed consent process.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2005-06 (Actual); Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W. Otto, Ph.D., Principal Investigator — Boston University; Mark H. Pollack, M.D., Principal Investigator — Rush University; Steven A. Safren, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Bay Cove Treatment Center, Boston, Massachusetts
  - Habit Management Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hearon BA, Calkins AW, Halperin DM, McHugh RK, Murray HW, Otto MW. Anxiety sensitivity and illicit sedative use among opiate-dependent women and men. Am J Drug Alcohol Abuse. 2011 Jan;37(1):43-7. doi: 10.3109/00952990.2010.535581. Epub 2010 Nov 19. PMID 21090958
- [Result] McHugh RK, Murray HW, Hearon BA, Pratt EM, Pollack MH, Safren SA, Otto MW. Predictors of dropout from psychosocial treatment in opioid-dependent outpatients. Am J Addict. 2013 Jan;22(1):18-22. doi: 10.1111/j.1521-0391.2013.00317.x. PMID 23398222
- [Result] McHugh RK, Weitzman M, Safren SA, Murray HW, Pollack MH, Otto MW. Sexual HIV risk behaviors in a treatment-refractory opioid-dependent sample. J Psychoactive Drugs. 2012 Jul-Aug;44(3):237-42. doi: 10.1080/02791072.2012.703507. PMID 23061323
- [Result] Otto MW, Hearon BA, McHugh RK, Calkins AW, Pratt E, Murray HW, Safren SA, Pollack MH. A randomized, controlled trial of the efficacy of an interoceptive exposure-based CBT for treatment-refractory outpatients with opioid dependence. J Psychoactive Drugs. 2014 Nov-Dec;46(5):402-11. doi: 10.1080/02791072.2014.960110. PMID 25364993

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via study flyers and postings or were referred to study staff by their substance abuse counselor.
Pre-assignment Details: 133 individuals were consented. Eleven dropped out prior to SCID administration. At the intake visit, 27 individuals were deemed ineligible. Of the 95 individuals who were eligible, 17 dropped out prior to randomization (7 were discharged, 2 declined treatment, and 8 were lost to contact). A total of 78 individuals were randomized to treatment.
Groups:
- Cognitive Behavioral Therapy: Cognitive Behavioral Therapy
  Cognitive Behavioral Therapy: 12 weekly sessions and 3 booster sessions of cognitive behavioral therapy
- Individual Drug Counseling: Individual Drug Counseling
  Individual Counseling: 12 weekly sessions and 3 booster sessions of individual counseling
Period: Completed Treatment
Arm/Group | Cognitive Behavioral Therapy | Individual Drug Counseling
Started | 41 | 37
Completed ASI at Midpoint | 35 | 29
Completed (Non-completion was operationalized as a failure to complete at least 12 of 15 treatment sessions.) | 34 | 26
Not Completed | 7 | 11
Not completed — Insufficient Treatment | 7 | 11
Period: Completed 2 Follow-Up Visits
Arm/Group | Cognitive Behavioral Therapy | Individual Drug Counseling
Started | 34 | 26
Completed ASI at Follow-Up #1 | 27 | 20
Completed ASI at Follow-Up #2 | 29 | 20
Completed | 29 | 20
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Population: Randomized sample
Groups:
- Cognitive Behavior Therapy: Psychosocial treatment with an individualized therapy emphasizing interoceptive exposure and training alternative responses to cues for drug use
- Individual Drug Counseling: Psychosocial treatment with individual drug counseling
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavior Therapy | Individual Drug Counseling | Total
Number analyzed (Participants) | 41 | 37 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (9.8) | 42.4 (10.0) | 42.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 23 | 20 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 36 | 34 | 70
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 11 | 25
  White | 27 | 26 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41 | 37 | 78

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Positive Toxicology Swabs for Illicit Substances
Description: The primary outcome assessment for this study was the percentage of oral toxicology swabs that were positive of illicit substances. Participants completed these swabs at each assessment point, as well as at each study therapy session. Toxicology swabs were supervised by study staff and used oral specimen collection to screen for opiates, methadone, cocaine, benzodiazepines, amphetamines, THC, and barbiturates.
Time Frame: Weekly assessments with summation over three time periods: baseline, treatment, and eight weeks of follow-up.
Population: Randomized participants
Measure: Mean (Standard Deviation); unit: percentage of positive toxicology screen
Arm/Group | Cognitive Behavioral Therapy | Individual Drug Counseling
Number analyzed (Participants) | 41 | 37
percentage of positive toxicology screen
  Baseline Period | 81.3 (24.3) | 79.1 (33.8)
  Treatment Period: number analyzed (Participants) | 37 | 31
  Treatment Period | 86.2 (18.7) | 82.3 (24.3)
  Follow-Up Period: number analyzed (Participants) | 34 | 29
  Follow-Up Period | 77.6 (27.4) | 74.8 (30.7)

2. Secondary Outcome: Addiction Severity Index (ASI) Drug Composite Index
Description: The composite score for drug use is determined by answers to 13 questions on the ASI: A/390 + B/390 + C/390 + D/390 + E/390 + F/390 + G/390 +H/390 + I/390 + J/390 + K/390 + L/52 + M/52. A single score is provided, with possible scores ranging from 0 to 1, with higher scores indicate greater drug use.
Time Frame: Baseline, Mid Treatment, Treatment Endpoint, Follow-up Evaluation 1, Follow-up Evaluation 2
Population: Randomized participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy | Individual Drug Counseling
Number analyzed (Participants) | 41 | 37
units on a scale
  Baseline: number analyzed (Participants) | 40 | 37
  Baseline | .23 (.09) | .21 (.12)
  Mid Treatment: number analyzed (Participants) | 35 | 29
  Mid Treatment | .20 (.07) | .16 (.10)
  Treatment Endpoint: number analyzed (Participants) | 34 | 26
  Treatment Endpoint | .17 (.09) | .18 (.13)
  Follow Up 1: number analyzed (Participants) | 27 | 20
  Follow Up 1 | .16 (.09) | .18 (.11)
  Follow-Up 2: number analyzed (Participants) | 29 | 20
  Follow-Up 2 | .16 (.12) | .16 (.12)

ADVERSE EVENTS:
Time Frame: Adverse event data were not formally collected. However, any informal report via a participant was recorded from the initial baseline session to the two follow-up assessments. All-cause mortality was not assessed.
Description: Because the study involved staff from both Boston University and Massachusetts General Hospital, participants signed a consent form for each institution. Subsequently, all serious adverse events (SAEs) were reported to the IRBs of both institutions. All SAEs were reported within 24 hours of discovery. SAE reports were collected in a non-systematic matter and all were judged by the investigators to be unrelated to the study procedures.
  Adverse events (AEs) were not assessed in this study.
Arm/Group | Cognitive Behavioral Therapy | Individual Drug Counseling
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 11/41 | 11/37
Other Adverse Events (participants affected / at risk) | 0/41 | 0/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Behavioral Therapy (N=41) | Individual Drug Counseling (N=37)
Foot Ulcer (General disorders) | 1 (1) | 0 (0) — A participant was hospitalized for a chronic foot ulcer problem. Hospitalization lasted for two weeks, but the participant still completed his study visits. The medical event was judged to be in no way related to the study procedures.
Ankle Sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Participant was partially hospitalized for a sprained left ankle. Hospitalization was required due to patient's perceived medical risk. This event was judged to be unrelated to study procedures.
Kidney infection (Renal and urinary disorders) | 1 (1) | 0 (0) — Participant was hospitalized due to a kidney infection secondary to an untreated urinary tract infection. This event was judged to be unrelated to study procedures.
Hairline fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Participant was admitted to the ER secondary to bruised ribs and hairline fracture secondary to falling from a chair.
Oversedation (Psychiatric disorders) | 0 (0) | 1 (1) — Participant was hospitalized secondary to "oversedation." Patient subsequently sought out inpatient detox, complaining of overprescription of a benzodiazepine medication and acute psychiatric symptoms.
Groin Injury (Renal and urinary disorders) | 1 (1) | 0 (0) — Participant was hospitalized due to problematic functioning in the patient's groin area.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Hospitalization due to pneumonia resulting from chronic condition that compromises immune functioning.
High Glucose Levels (Endocrine disorders) | 0 (0) | 1 (1) — Hospitalization due to extremely high glucose levels resulting from diabetes.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Participant was hospitalized for four days due to pneumonia, inflamed intestines, and high blood pressure (as per patient report). Investigators learned about the SAE after patient has been discharged.
Respiratory Problems (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Hospitalization due to low blood pressure and respiratory problems.
Detoxification (Psychiatric disorders) | 1 (1) | 0 (0) — Participant reported being admitted to a residential substance abuse treatment facility for detoxification. The patient remained at the facility for 30 days. The admission to the facility occurred prior to randomization to treatment condition.
Depression (Psychiatric disorders) | 1 (1) | 0 (0) — Inpatient psychiatry hospitalization for six days due to symptoms of depression. Patient denied suicidal ideation, and stated that hospitalization was required for emergency medication management.
Blood Clot (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Hospitalization for five days due to formation of a blood clot around the central artery, where a central IV had previously been placed. Patient was treated by hospital staff with prescribed self-injection and a blood thinner.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Hospitalization for seven days due to a bout of pneumonia.
Hospitalization for Chronic Health Concerns (General disorders) | 1 (1) | 0 (0) — Hospitalization for four days. Participant had chronic health concerns and completed the active treatment phase of the study and had been discharged from the clinic before hospitalization. This SAE was unrelated to study procedures.
Infection (General disorders) | 0 (0) | 1 (1) — Hospitalization for two to three days for an infection and unspecified chronic health problems. Participant resumed and completed study procedures upon discharge from the hospital. This event was unrelated to study procedures.
Detoxification (Psychiatric disorders) | 0 (0) | 1 (1) — Participant voluntarily entered an inpatient unit for five days for the detoxification of benzodiazepines. Participant resumed and completed study procedures upon discharge from the hospital. This event was unrelated to study procedures.
Detoxification (Psychiatric disorders) | 0 (0) | 1 (1) — Participant was hospitalized for detoxification and mental health problems. This participant was subsequently discharged from the methadone clinic and did not complete study procedures. This event was unrelated to study procedures.
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1) — Participant reported losing housing, and reported suicidal ideation to a (non-study) counselor to obtain emergency housing. Participant was at this unit for several days, yet came to the methadone clinic as part of scheduled study involvement.
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1) — Participant reported serious psychological distress to study staff. After assessing suicidal ideation, it was decided that this situation warranted intervention.The participant was then independently assessed and hospitalization by clinic staff.
Detoxification (Psychiatric disorders) | 0 (0) | 1 (1) — Participant voluntarily entered an inpatient detoxification unit for the detoxification of heroin and benzodiazepines. Upon discharge from the detoxification facility, the participant resumed regular study involvement and completed study procedures.
Detoxification (Psychiatric disorders) | 1 (1) | 0 (0) — Participant voluntarily entered an inpatient unit for 5 days for the detoxification of benzodiazepines. Upon discharge from the detoxification facility, the participant resumed regular dosing at the methadone clinic and resumed study procedures.
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1) — The investigators were notified that a participant was hospitalized again for suicidal ideation. The clinic staff independently assessed the patient and deemed that hospitalization was necessary.
Detoxification (Psychiatric disorders) | 0 (0) | 1 (1) — Participant voluntarily entered an inpatient detoxification unit. Upon discharge from the detoxification facility, the participant resumed regular study involvement.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Participant was hospitalized for 7 days for pneumonia. This participant has a history of chronic health problems, which worsened to the point that IV antibiotics were needed. Participant resumed dosing at the clinic and resumed study procedures.
Stab Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Participant was hospitalized for five days for various medical problems related to a stab wound, including several blood transfusions. Participant resumed dosing at the clinic and resumed study procedures.
Kidney Stone (Renal and urinary disorders) | 1 (1) | 0 (0) — Participant was hospitalized for several days for a kidney stone. Participant was released and resumed dosing at the clinic and resumed study procedures.
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Participant hospitalized for dehydration. Following discharged, participant resumed dosing at the clinic and continued with study procedures.
Wound Treatment (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Participant was hospitalized overnight for 3 days. Participant was beaten over the head and received treatment for his wounds at this hospital. Participant resumed dosing at the clinic and continued study procedures.
Hospitalization for Chronic Health Concerns (General disorders) | 0 (0) | 1 (1) — Hospitalization for four days. Participant had chronic health concerns and completed the active treatment phase of the study and had been discharged from the clinic before hospitalization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes